CLINICAL TRIAL: NCT02187666
Title: National Neurosurgical and Orthopedic Optimum Care Continuum Spine Registry Exposure for Various Implants/Products
Brief Title: NOC2 Spine Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: DC2 Healthcare (Industry)
Collaborators: National Neurosurgical and Orthopedic Optimum Care Continuum (NOC2) (Unknown); National Research Independent Operations Management (Other)
Responsible Party: Sponsor
Other Study IDs: NOC 1001
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Spinal Disease
Keywords: Cervical; Lumbar; Spine; Spinal Disease
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lumbar: Patients undergoing lumbar spinal surgery
- Cervical: Patients undergoing cervical spine surgery

SUMMARY:
The primary objective of the Spine Registry is to enhance the understanding of spinal disease and treatment of spinal disease with the goal of guiding treatment options.

DETAILED DESCRIPTION:
This study will enhance the understanding of the variability, progression and treatment of spinal disease with the ultimate goal of better guiding and assessing therapeutic intervention. Researchers will collect complications and safety following cervical and lumbar surgeries to determine best options for patients. Prospective reports will be collected on patients undergoing lumbar or cervical spinal surgery. Patients will be enrolled in registry after signing informed consent. Data will be collected at various time points. The registry will serve as a database of cervical and lumbar surgeries in which retrospective analysis and exploratory analysis of specific research questions can be answered.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lumbar or cervical surgery
* Understand and sign informed consent

Exclusion Criteria:

* There are no specific exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 10,000 patients undergoing lumbar or cervical surgery will be screened to decide whether they meet the inclusion and exclusion criteria of the study/patient registry. Patients who meet the study criteria will be informed by the investigator and should read the 'patient information' document. Patients must give their written informed consent to be enrolled into this study.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2011-12; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analogue Scale (VAS) from baseline at 4 weeks | baseline and 4 weeks after surgery
  Pain intensity scale taken at baseline and 4 weeks after surgery
Change in Visual Analogue Scale (VAS) from baseline at 3 months | baseline and 3 months after surgery
  Pain intensity scale taken at baseline and 3 months after surgery
Change in Visual Analogue Scale (VAS) from baseline at 6 months | baseline and 6 months after surgery
  Pain intensity scale taken at baseline and 6 months after surgery
Change in Visual Analogue Scale (VAS) from baseline at 12 months | baseline and 12 months after surgery
  Pain intensity scale taken at baseline and 12 months after surgery
Change in Visual Analogue Scale (VAS) from baseline at 24 months | baseline and 24 months after surgery
  Pain intensity scale taken at baseline and 24 months after surgery

SECONDARY OUTCOMES:
Change from baseline in Oswestry Disability index at 4 weeks | baseline and 4 weeks after surgery
  Assesses impact of disability in terms of activities of daily living. To be taken at baseline and 4 weeks after surgery.
Fusion at 6 months | 6 months post-op
Length of hospital stay | one to three days following surgery
  Date of discharge will be recorded, an average of one to three days
Revision surgery within 30 days | 30 days after surgery
Return to work | 4 weeks after surgery
  Time off of work and whether patient returned restricted or unrestricted
Return to normal/usual activity | 4 weeks after surgery
  Time between surgery and resuming normal activity for patient
Complications | 24 hours after surgery
Change from baseline in Oswestry Disability index at 3 months | baseline and 3 months after surgery
  Assesses impact of disability in terms of activities of daily living. To be taken at baseline and 3 months after surgery.
Change from baseline in Oswestry Disability index at 6 months | baseline and 6 months after surgery
  Assesses impact of disability in terms of activities of daily living. To be taken at baseline and 6 months after surgery.
Change from baseline in Oswestry Disability index at 12 months | baseline and 12 months after surgery
  Assesses impact of disability in terms of activities of daily living. To be taken at baseline and 12 months after surgery.
Change from baseline in Oswestry Disability index at 24 months | baseline and 24 months after surgery
  Assesses impact of disability in terms of activities of daily living. To be taken at baseline and 24 months after surgery.
Return to work | 3 months after surgery
  Time off of work and whether patient returned restricted or unrestricted
Return to work | 6 months after surgery
  Time off of work and whether patient returned restricted or unrestricted
Return to work | 12 months after surgery
  Time off of work and whether patient returned restricted or unrestricted
Return to work | 24 months after surgery
  Time off of work and whether patient returned restricted or unrestricted
Return to normal/usual activity | 3 months after surgery
  Time between surgery and resuming normal activity for patient
Return to normal/usual activity | 6 months after surgery
  Time between surgery and resuming normal activity for patient
Return to normal/usual activity | 12 months after surgery
  Time between surgery and resuming normal activity for patient
Return to normal/usual activity | 24 months after surgery
  Time between surgery and resuming normal activity for patient
Complications | 4 weeks after surgery
Complications | 3 months after surgery
Complications | 6 months after surgery
Complications | 12 months after surgery
Complications | 24 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- DC2 Healthcare, Nashville, Tennessee, United States

REFERENCES:
- See also: DC2 Healthcare — http://www.dc2healthcare.com
- See also: NRIOM — http://www.nriom.com/